CLINICAL TRIAL: NCT01027182
Title: Comparison of Concentration-time Course of Plasma and Intracellular Raltegravir in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Changi General Hospital (Other)
Collaborators: National University Hospital, Singapore (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Professor Edmund Lee, Changi General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: RAL
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2010-03

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Raltegravir (No Intervention)
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — One 400mg tablet on day 1.
  Other Names: ISENTRESS, 400mg

SUMMARY:
The investigators hypothesize that the concentration-time profile of raltegravir is different in cells than that in plasma. Intracellular raltegravir concentrations may be higher and its half-life longer than in plasma. This may explain the efficacy of raltegravir despite variable plasma concentrations.

DETAILED DESCRIPTION:
In less than 15 years, human immunodeficiency virus (HIV) infection has reached the level of a pandemic, and acquired immunodeficiency syndrome (AIDS) has been reported in over 190 countries. By the end of 2001, more than 30 million people were infected with HIV worldwide, with approximately one million of those infected residing in North America and one million residing in Europe.

Significant advances have been made in the treatment of HIV disease. The nucleoside reverse transcriptase inhibitors provided the earliest therapeutic intervention for HIV infection. This class of antiretroviral agents interferes with the replication of HIV by competitive inhibition of the HIV reverse transcriptase enzyme and by chain termination of new HIV DNA into which the nucleoside analogue has been incorporated. Subsequent development of other potent drug classes, such as non nucleoside reverse transcriptase inhibitors and protease inhibitors, has made possible the use of multidrug, multiclass regimens that can achieve durable suppression of HIV replication. However, extensive resistance has developed to these classes of drugs, necessitating the development of other potent classes of antiretroviral therapy.

The integrase inhibitors are a new class of antiretroviral drugs. They inhibit the catalytic activity of HIV integrase, an HIV encoded enzyme that is required for viral replication. Inhibition of integrase prevents the covalent insertion, or integration, of unintegrated linear HIV DNA into the host cell genome preventing the formation of the HIV provirus. The provirus is required to direct the production of progeny virus, so inhibiting integration prevents propagation of the viral infection.

Raltegravir (RAL) is a newly approved HIV integrase inhibitor. It is approved in salvage regimens(Merck &Co Inc. 2007) and shows promise in first line therapy. Raltegravir is potent in vitro; concentrations of 31 ± 20 nM resulted in 95% inhibition (EC95) of viral spread (relative to an untreated virus-infected culture) in human T-lymphoid cell cultures infected with the cell-line adapted HIV-1 variant H9IIIB. In addition, raltegravir at concentrations of 6 to 50 nM resulted in 95% inhibition of viral spread in cultures of mitogen-activated human peripheral blood mononuclear cells infected with diverse, primary clinical isolates of HIV-1, including isolates resistant to reverse transcriptase inhibitors and protease inhibitors.

RAL plasma concentrations are highly variable even after controlling for food intake and UGT1A1*28 polymorphisms. Despite this variability, RAL remains efficacious and studies have shown little correlation between various RAL pharmacokinetic parameters and efficacy(Wenning, Hwang et al. 2008). This suggests that although RAL exposure may be important, plasma concentrations may not the best marker of RAL exposure.

RAL exerts its effects in the HIV-infected cells where it inhibits the HIV integrase. Therefore intracellular concentrations should correlate with efficacy much more than plasma concentrations. It is possible that RAL could accumulate inside HIV-infected cells or that intracellular concentrations could be less variable, explaining the sustained efficacy of RAL despite variable plasma concentrations. Intracellular half-life could also be longer than the relatively short plasma half-life. This information could be used to justify once daily administration of RAL, just as zidovudine dosing was changed from five times to twice daily because intracellular zidovudine triphosphate had a much longer half-life than plasma zidovudine(Barry, Khoo et al. 1996).

Measurement of intracellular raltegravir could also aid in therapeutic drug monitoring and assessing drug-drug interactions. For example, rifampin reduces plasma concentration of RAL by almost 50%(Wenning, Hanley et al. 2009). However, dose increases may not be necessary if intracellular concentrations are maintained, as is thought to be true for zidovudine after rifampin co-administration.

To our knowledge, there has been no data on intracellular raltegravir. We therefore aim to measure the time course of RAL intracellular concentrations after a single dose in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 18 to 30 kg/m2, inclusive. BMI = weight (kg)/ [height (m)]2 and weigh at least 50kg.
* Non-smoking or smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 3 months prior to selection.
* Women of childbearing potential (WOCBP) must not be nursing or pregnant.
* Women of childbearing potential (have not been postmenopausal for at least 2 years nor undergone total hysterectomy) must have a negative serum Beta-HCG test performed at screening.
* Female subjects who are not of reproductive potential (have been postmenopausal for at least 2 years or undergone total hysterectomy) or whose male partner has undergone successful vasectomy with resultant azoospermia or has azoospermia for any other reason, are eligible without requiring the use of contraception. Documentation of menopause, sterilization (total hysterectomy or vasectomy) and azoospermia must be provided to study personnel at time of screening.
* Both male and female study volunteers of reproductive potential must agree not to participate in a conception process (i.e., active attempt to become pregnant or to impregnate via sperm donation or in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, the female study volunteer/male partner must use a form of contraception as specified below while receiving protocol-specified medication(s) and for 7 days after stopping the medication(s). Male study volunteers will be required to use a barrier method for at least 7 days after completion of the study.

Exclusion Criteria:

* History or current evidence of any significant acute or chronic medical illness that, within the investigator's discretion, would interfere with the conduct or interpretation of the study.
* Proven or suspected acute hepatitis at the time of study entry.
* Current or recent (within 3 months) gastrointestinal disease which would interfere with the conduct or interpretation of the study.
* Any major surgery within 8 weeks of enrollment. Any gastrointestinal surgery that could impact upon the absorption of study drug.
* Donation of blood or plasma within 60 days of screening.
* Inability to tolerate oral medication.
* Inability to tolerate venepuncture and/or absence of secure venous access.
* Inability to give informed consent voluntarily before the first trial-related activity.
* Known or suspected HIV infection or chronic HBV or HCV infection
* Known active drug or alcohol abuse, which in the opinion of the investigator makes study participation to completion unlikely.
* Any other significant medical, psychiatric and/or social issue as determined by the Investigator that would compromise subject's safety and/or compliance with trial procedures.
* Subjects with AST, ALT or total bilirubin above the upper limit of normal.
* Haemoglobin < 10.9 g/dL, and platelet count < 125,000/mm3.
* Creatinine clearance <60 ml/min
* Lipase or pancreatic amylase >1.1x ULN
* Fasting triglyceride >300 mg/dL.
* Absolute Neutrophil Count (ANC) <1300/mm3
* Serum creatinine grade 1 or greater (≥ 1.1 x upper limit of laboratory normal range [ULN])
* Any other clinically significant screening lab abnormality (as determined by the investigator)
* Exposure to any investigational drug (excluding raltegravir) within 90 days of enrollment and throughout the study.
* Any previous clinically significant allergy or hypersensitivity or intolerance to raltegravir or any other ingredient of the tablets.
* Use of any agent, within 2 weeks of dosing, that is known to induce or inhibit drug metabolizing enzymes.
* Use of concomitant medication, including investigational, prescription, and any over-the-counter drugs and dietary supplements with the following exceptions, aspirin, acetaminophen, chlorpheniramine, daily multivitamins, mineral supplements and hormonal oral contraceptives. Concomitant medication other than those listed above must have been discontinued within 14 days of study entry.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To determine the time course and half-life of intracellular raltegravir after a single dose, and compare with plasma concentrations. | 3 months

SECONDARY OUTCOMES:
To develop analytical methods to measure intracellular raltegravir using liquid chromatography / mass spectrometry (LCMS). | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Edmund JD Lee, Professor, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Barry MG, Khoo SH, Veal GJ, Hoggard PG, Gibbons SE, Wilkins EG, Williams O, Breckenridge AM, Back DJ. The effect of zidovudine dose on the formation of intracellular phosphorylated metabolites. AIDS. 1996 Oct;10(12):1361-7. doi: 10.1097/00002030-199610000-00008. PMID 8902065
- [Background] Long MC, Bennetto-Hood C, Acosta EP. A sensitive HPLC-MS-MS method for the determination of raltegravir in human plasma. J Chromatogr B Analyt Technol Biomed Life Sci. 2008 May 15;867(2):165-71. doi: 10.1016/j.jchromb.2008.03.022. Epub 2008 Apr 1. PMID 18430616
- [Background] Ter Heine R, Hillebrand MJ, Rosing H, van Gorp EC, Mulder JW, Beijnen JH, Huitema AD. Quantification of the HIV-integrase inhibitor raltegravir and detection of its main metabolite in human plasma, dried blood spots and peripheral blood mononuclear cell lysate by means of high-performance liquid chromatography tandem mass spectrometry. J Pharm Biomed Anal. 2009 Feb 20;49(2):451-8. doi: 10.1016/j.jpba.2008.11.025. Epub 2008 Nov 27. PMID 19128911
- [Background] Wenning LA, Hanley WD, Brainard DM, Petry AS, Ghosh K, Jin B, Mangin E, Marbury TC, Berg JK, Chodakewitz JA, Stone JA, Gottesdiener KM, Wagner JA, Iwamoto M. Effect of rifampin, a potent inducer of drug-metabolizing enzymes, on the pharmacokinetics of raltegravir. Antimicrob Agents Chemother. 2009 Jul;53(7):2852-6. doi: 10.1128/AAC.01468-08. Epub 2009 May 11. PMID 19433563
- [Background] Wenning, L. A., E. Hwang, et al. (2008). Pharmacokinetic/Pharmacodynamic (PK/PD) Analyses for Raltegravir (RAL) in Phase III Studies in Treatment Experienced HIV- Infected Patients Following 48 Weeks of Treatment. ICAAC. Washington DC, USA
- [Background] Merck &Co Inc. (2007). Isentress (raltegravir) tablets. FDA approved label.